CLINICAL TRIAL: NCT07052851
Title: Performance of CCoat Intra-Articular Injections in Mild to Moderate Knee Osteoarthritis: A Prospective, Randomized, Double-Blind, Multi-center Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lipo-Sphere (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLD0001465
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant, Investigator and sponsor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCoat, Liposphere Ltd. (Experimental): CCoat is indicated for patients with mild to moderate OA of the knee. a single IA injection of 4 ml CCoat
  Interventions: Device: CCoat, Liposphere Ltd
- Synvisc-One® (hylan G-F 20), (Active Comparator): intra-articular injection, 6 mL single-dose syringe, Genzyme Corporation
  Interventions: Device: Synvisc-One® (hylan G-F 20)

INTERVENTIONS:
Device: CCoat, Liposphere Ltd — a single IA injection of 4 ml CCoat
  Arms: CCoat, Liposphere Ltd.
Device: Synvisc-One® (hylan G-F 20) — Group 2 (Active Comparator): a single IA Synvisc-One® (hylan G-F 20) of 6 mL, Genzyme Corporation
  Arms: Synvisc-One® (hylan G-F 20),

SUMMARY:
Performance of CCoat Intra-Articular Injections in Mild to Moderate Knee Osteoarthritis: A Prospective, Randomized, Double-Blind, Multi-center Trial

DETAILED DESCRIPTION:
The study aims to evaluate the performance of a single intra-articular injection of CCoat in patients with mild to moderate knee osteoarthritis over 26 weeks. Intra-articular injections are widely used for their localized efficacy and reduced systemic toxicity compared to oral treatments. Current treatments, including corticosteroids and hyaluronic acid, have limitations such as short-term effects and potential cartilage damage [1],[2],[3],[4]. Platelet-rich plasma (PRP) and mesenchymal stem cells (MSCs) offer promise but require further validation [5],[6],[7]. CCoat, a liposomal boundary lubricant, provides a novel approach by coating cartilage surfaces to reduce wear, offering mechanical protection without altering synovial fluid properties.

CCoat is a new intra-articular (IA) injectable joint lubricant for patients suffering from mild to moderate knee osteoarthritis (OA), developed by Liposphere LTD. CCoat is a liposomal boundary lubricant that coats the cartilage surface and temporarily protects it from further damage and degradation.

The performance and safety of CCoat device over 26 weeks is being evaluated in another multi-center, prospective, placebo controlled, randomized, double- blinded clinical study in 150 patients with mild to moderate OA of the knee (per study protocol # CLD0000616). As this study is ongoing, there is no currently available data related to the performance of the device. With regards to the CCoat's safety, in the interim analysis no safety concerns were raised.

This clinical investigation aims to further confirm the performance of CCoat when used as intended for the treatment of mild to moderate knee osteoarthritis (OA) in a larger patient population group, in comparison to a marketed hyaluronic acid product. This study is critical to further confirm the benefit-risk profile of the CCoat device as a valid therapeutic option for knee OA treatment, which remains a significant unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated the informed consent form (ICF).
2. Age ≥18 years.
3. Participants must have a KOOS Pain subscale score of 25≤75 in the index knee over the last week before screening.

   * Minimum baseline severity: At least two items in the KOOS Pain Subscale must be scored as moderate or worse (score 2-4 on the 0-4 scale).
   * Pain consistency: Subjects must have experienced knee pain on most days in the past month to exclude acute or transient cases.
4. Participants must have a KOOS Symptoms subscale score of 30≤ 75 in the index knee over the last week before screening. Subjects must report at least moderate severity (score ≥2) in at least one of the following:

   * Knee stiffness in the morning
   * Knee stiffness after sitting/resting
   * Swelling in the knee
5. Degenerative changes in the index knee that can be categorized as grade II -III- Kellgren Lawrence based upon standing anterior- posterior and lateral radiographs of the knee.
6. Body Mass Index (BMI) between 18.5 kg/m2 and 38 kg/m2
7. A negative urine pregnancy test female patient with childbearing potential at Visit 1 prior to intra-articular injection of CCoat.
8. If female, the subject must be either postmenopausal, OR permanently surgically sterile OR for women of childbearing potential using at least 2 methods of birth control that are effective from at least 30 days before Visit 1 through visit 26 w (26 weeks post injection).
9. Are willing or able to comply with the procedures required in this protocol.

Exclusion Criteria:

1. Osteoarthritis of the index knee graded 4 according to the Kellgren- Lawrence Grading.
2. History of significant knee trauma or previous surgery of the intended study knee within the last 3 months preceding the screening.
3. KOOS Pain subscale score of ≤25 or >75 in the index knee.
4. Pain in the contra lateral knee: KOOS Pain subscale score of ≤75.
5. Intra-articular injection to the intended study knee within 3 months before screening.
6. Significant instability of the index knee.
7. Malalignment of more than 10 degrees varus OR 10 degrees valgus according to standing X-ray.
8. Intake of chronic pain medications (especially opioid pain relievers) without an option to pause for the period of the study.
9. History of Psoriatic Arthritis, Rheumatoid Arthritis, or any other inflammatory condition associated with arthritis.
10. Wound in the area of the index knee.
11. Any known tumor of the index knee.
12. Any known history of intra-articular or osseous infection of the index knee.
13. Any evidence of active infection anywhere in the body.
14. Any known systemic cartilage and/or bone disorder, such as but not limited to, chondrodysplasia or osteogenesis imperfecta.
15. Active malignancies, excluding BCC.
16. Chemotherapy and/or radiation in the past 12 months.
17. Known history of a severe allergic reactions.
18. Patient who is pregnant or intends to become pregnant during the study.
19. Breastfeeding female patients.
20. History of any significant systemic disease, such as but not limited to: hepatitis and coagulopathies.
21. Immunosuppressives, anti-coagulants.
22. A known substance or alcohol abuse.
23. Participation in other clinical trials within 60 days to before the study or concurrent with the study.
24. Known insulin dependent diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Knee injury and Osteoarthritis Outcome Score (KOOS) Pain score at 12 weeks | Time Frame: Day 0, up to week 12
  The change in KOOS Pain score from baseline to 12 weeks visit will be compared between the treatment groups using a repeated measures analysis of covariance (ANCOVA, SAS® MIXED procedure). The model will include the following fixed effects: treatment group, visit, treatment group by visit interaction with Baseline KOOS Pain, K/L grade, and center entered as covariates. The principal statistical analysis will be a comparison between the treatment groups, derived from the visit by treatment group interaction term from the model. The adjusted mean change from baseline in KOOS Pain scores at 12 weeks post treatment initiation will be estimated from the model (LS Means) interaction term for each group as well as the difference between the adjusted means and presented together with 95% Confidence Intervals (CI's).

SECONDARY OUTCOMES:
The secondary objective is to assess change from baseline to 2 and 12 weeks in KOOS Symptoms and ADL scores. | baseline to 2 and 12 weeks in KOOS Symptoms and ADL scores.
  * Change from baseline in Knee injury and Osteoarthritis Outcome Score (KOOS) Symptoms score at 12 weeks - [Time Frame: Day 0, up to week 12]
  * Change from baseline in Knee injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living (ADL) score at 12 weeks - [Time Frame: Day 0, up to week 12]
  * Change from baseline in Knee injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QoL) score at 12 weeks - [Time Frame: Day 0, up to week 12]